CLINICAL TRIAL: NCT03351556
Title: Optimizing the Efficiency and Implementation of Cash Transfers to Improve Adherence to Antiretroviral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Rasello (Industry); Health for a Prosperous Nation (Other); Management and Development for Health in Tanzania (Unknown)
Responsible Party: Principal Investigator, Sandra McCoy, PI, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH112432-01A1 (NIH); R01MH112432-01A1 (NIH)
Record Dates: First submitted 2017-11-19; First posted 2017-11-24 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: HIV/AIDS; Adherence, Medication; Adherence, Patient
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the cash transfer arms will be masked to the knowledge that there are two cash value arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comparison Arm (No Intervention): Participants in the comparison group will receive the standard HIV primary care services according to Tanzania's National Guidelines for the Management of HIV and AIDS.
- Active Intervention 1 (Experimental): Participants will receive the standard HIV primary care services according to Tanzania's National Guidelines for the Management of HIV and AIDS plus the opportunity to earn 10,000 TZS/month (~$4.50) for up to 6 months conditional on visit attendance.
  Interventions: Behavioral: Active Arm 1
- Active Intervention 2 (Experimental): Participants will receive the standard HIV primary care services according to Tanzania's National Guidelines for the Management of HIV and AIDS plus the opportunity to earn 22,500 TZS/month (~$10.00) for up to 6 months conditional on visit attendance.
  Interventions: Behavioral: Active Arm 2

INTERVENTIONS:
Behavioral: Active Arm 1 — Participants in this arm will receive the standard HIV primary care services according to Tanzania's National Guidelines for the Management of HIV and AIDS plus the opportunity to earn 10,000 TZS/month conditional on visit attendance.
  Arms: Active Intervention 1
Behavioral: Active Arm 2 — Participants in this arm will receive the standard HIV primary care services according to Tanzania's National Guidelines for the Management of HIV and AIDS plus the opportunity to earn 22,500 TZS/month conditional on visit attendance.
  Arms: Active Intervention 2

SUMMARY:
1. Determine the "dose-response" relationship between a cash transfer amount and HIV viral suppression at 6 months
2. Identify the most effective cash transfer size to increase the proportion of people living with HIV infection (PLHIV) retained in care and with suppressed viral load (<1000 copies/ml) after 6 months. (This amount will be further evaluated in a cluster randomized trial in Phase 2).

DETAILED DESCRIPTION:
Participants in the control group will receive the standard HIV primary care services according to Tanzania's National Guidelines for the Management of HIV and AIDS.

The study has two active intervention arms:

1. The opportunity to earn 10,000 TZS/month (~$4.50) for up to 6 months conditional on visit attendance, and
2. The opportunity to earn 22,500 TZS/month (~$10.00) for up to 6 months conditional on visit attendance

In both intervention arms, cash transfers will be delivered a maximum of once monthly, spaced ≥28 days apart, for up to six months and delivered via an automatic mobile money system linked to a biometric identification system.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Living with HIV infection
* Initiated antiretroviral therapy ≤1 month prior to enrollment in the study

Exclusion Criteria:

- Participants who do no provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HIV viral suppression at 6 months | 6 months
  <1000 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I McCoy, PhD, Principal Investigator — University of California, Berkeley; Prosper Njau, MD, MPH, Principal Investigator — Health for a Prosperous Nation and Ministry of Health, Community Development, Gender, Elderly, and Children
Locations (4):
- Tanzania (4):
  - Kahama Hospital, Kahama, Shinyanga
  - Kagongwa Health Center, Shinyanga, Shinyanga
  - Kambarage Health Center, Shinyanga, Shinyanga
  - Shinyanga Regional Referral Hospital, Shinyanga, Shinyanga

REFERENCES:
- [Derived] Winters S, Sabasaba A, Fahey CA, Packel L, Katabaro E, Ndungile Y, Njau PF, McCoy SI. Increased prevalence of depression and anxiety among adults initiating antiretroviral therapy during the COVID-19 pandemic in Shinyanga region, Tanzania. AIDS Res Ther. 2023 Jun 10;20(1):36. doi: 10.1186/s12981-023-00534-y. PMID 37301833
- [Derived] Packel L, Fahey C, Kalinjila A, Mnyippembe A, Njau P, McCoy SI. Preparing a financial incentive program to improve retention in HIV care and viral suppression for scale: using an implementation science framework to evaluate an mHealth system in Tanzania. Implement Sci Commun. 2021 Sep 23;2(1):109. doi: 10.1186/s43058-021-00214-w. PMID 34556176
- [Derived] Fahey CA, Njau PF, Katabaro E, Mfaume RS, Ulenga N, Mwenda N, Bradshaw PT, Dow WH, Padian NS, Jewell NP, McCoy SI. Financial incentives to promote retention in care and viral suppression in adults with HIV initiating antiretroviral therapy in Tanzania: a three-arm randomised controlled trial. Lancet HIV. 2020 Nov;7(11):e762-e771. doi: 10.1016/S2352-3018(20)30230-7. Epub 2020 Sep 3. PMID 32891234